CLINICAL TRIAL: NCT05509192
Title: Intubation Conditions Achieved With Rapid Co-administration of Rocuronium and Propofol Versus Classical Induction: A Prospective Randomized and Blind Trial
Brief Title: Intubation Conditions Achieved With Rapid Co-administration of Rocuronium and Propofol Versus Classical Induction
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Lauren Nakazawa, Assistant Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HSC-MS-22-0495
Record Dates: First submitted 2022-08-16; First posted 2022-08-22 (Actual); Results first posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-01

CONDITIONS: Anesthesia

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- MTPI group (Experimental)
  Interventions: Drug: MTPI
- Classic Induction group (Active Comparator)
  Interventions: Drug: Classic Induction

INTERVENTIONS:
Drug: MTPI — Patients from both study groups will receive premedication in the usual fashion, typically 0-2 mg of IV midazolam at the discretion of the care team. Patients in both study groups will receive 1 mg/kg of lidocaine intravenously, followed by an opioid such as fentanyl (1-2 mcg/kg), prior to administration of induction drugs. Patients assigned to MTPI will then be given rocuronium (0.6mg/kg), followed by propofol intravenously as a single bolus within 10 seconds. A typical propofol bolus for induction ranges from 1-2mg/kg, depending on the patient's age, medical history, and co-morbidities. Propofol dosing will be at the discretion of the care team. Patients will count down from one hundred. Once apnea occurs, as indicated by a lack of respiratory effort, the eyes will be taped, and intubation with C-MAC (Karl Storz 8403ZX, Tuttlingen, Germany) is initiated.
  Arms: MTPI group
Drug: Classic Induction — Patients assigned to CI will be induced as per routine care using lidocaine 1 mg/kg, an opioid such a fentanyl (1-2 mcg/kg), propofol 1-2 mg/kg, and rocuronium 0.6 mg/kg, and the intubation will be performed with a C-MAC. Patients will also count down from one hundred. The medications used for induction of anesthesia in both arms of the study are those used for routine anesthesia care. In both study arms, dosing of medications for induction of anesthesia is standardized (lidocaine 1 mg/kg, fentanyl 1-2 mcg/kg, propofol 1-2 mg/kg, and rocuronium 0.6 mg/kg). The only difference between the two arms will be the timing of the medication administration, and the order in which medications are administered. The documentation of induction and intubation will be the same as that of the MTPI group. Vital signs and other parameters will continuously be recorded in the intraoperative record. Emergence and extubation are not protocolized.
  Arms: Classic Induction group

SUMMARY:
The purpose of this study is to assess and compare the conditions for tracheal intubation obtained with Modified Time Principle Induction (MTPI) and that obtained with classic induction (CI). This study will compare the efficiency of tracheal intubation with the two induction techniques, as well as evaluate for potential adverse events.

ELIGIBILITY:
Inclusion Criteria:

* BMI >30 kg/M2 or Mallampati class III or IV
* Requiring general anesthesia and endotracheal intubation

Exclusion Criteria:

* Acute and chronic respiratory disorders, including Chronic obstructive pulmonary disease (COPD) and asthma
* American Society of Anesthesiologists (ASA) physical status classification > III
* Emergency surgery
* Induction requiring cricoid pressure
* Patients requiring awake intubation
* Pregnant women
* Patients who require an induction dose of propofol less than 1 mg/kg
* Untreated ischemic heart disease
* Contraindication to mask ventilation
* Allergy to propofol, rocuronium, or Sugammadex
* Induction requiring succinylcholine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2022-08-17 (Actual); Primary Completion 2025-01-24 (Actual); Study Completion 2025-01-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lauren M Nakazawa, MD, MBA, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | MTPI Group | Classic Induction Group
Started | 77 | 77
Received Intervention | 77 | 74
Completed | 64 | 68
Not Completed | 13 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MTPI Group | Classic Induction Group | Total
Number analyzed (Participants) | 64 | 68 | 132
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.7 (15.3) | 46.6 (15.0) | 47.2 (15.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 40 | 77
  Male | 27 | 28 | 55
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
American Society of Anesthesiology (ASA) Classification [Count of Participants; unit: Participants] — ASA Physical Status Classification System - The purpose of the system is to assess and communicate a patient's pre-anesthesia medical co-morbidities.
  ASA I :A normal healthy patient ASA II :A patient with mild systemic disease ASA III: A patient with severe systemic disease ASA IV: A patient with severe systemic disease that is a constant threat to life
  Participants
    ASA I: A normal healthy patient | 2 | 5 | 7
    ASA II: A patient with mild systemic disease | 22 | 25 | 47
    ASA III: A patient with severe systemic disease | 39 | 38 | 77
    ASA IV: A patient with severe systemic disease that is a constant threat to life | 1 | 0 | 1
Mallampati class [Count of Participants; unit: Participants] — The Mallampati score assesses the relative size of the tongue base in relation to the oropharyngeal opening to predict potential airway difficulty. It is assessed categorically as follows:
  Class I: Full view of soft palate, uvula, and tonsillar pillars Class II: Soft palate and uvula visible, pillars obscured Class III: Soft palate and uvula base visible Class IV: Visualization restricted to the hard palate
  Participants
    Class I | 13 | 15 | 28
    Class II | 29 | 26 | 55
    Class III | 17 | 19 | 36
    Class IV | 4 | 5 | 9
    Unknown | 1 | 3 | 4
Patients with both BMI ≥ 30 and Mallampati class ≥ 3 [Count of Participants; unit: Participants] | 19 | 20 | 39
Providers' training levels [Count of Participants; unit: Participants]
  Attending Anesthesiologists | 8 | 14 | 22
  Anesthesia assistants | 14 | 9 | 23
  Anesthesia residents | 42 | 45 | 87
Height [Mean (Standard Deviation); unit: centimeters] | 169.8 (11.3) | 169.6 (10.6) | 169.7 (10.9)
Weight [Mean (Standard Deviation); unit: Kilograms] | 110.8 (28.2) | 107.4 (25.6) | 109.0 (26.8)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 38.2 (8.0) | 36.6 (7.9) | 37.7 (8.0)

OUTCOME MEASURES:

1. Primary Outcome: The Total Time Between Laryngoscope Insertion Into Mouth and the Onset of Ventilation After Tracheal Intubation
Time Frame: Between laryngoscope insertion to onset of ventilation (less than 7 minutes)
Measure: Median (Inter-Quartile Range); unit: seconds
Arm/Group | MTPI Group | Classic Induction Group
Number analyzed (Participants) | 64 | 68
seconds | 30.0 [22.0 to 41.5] | 33.0 [28.0 to 50.0]

2. Secondary Outcome: Number of Participants for Whom Tracheal Intubations Were Successful on the First Attempt
Time Frame: after 5 minutes of successful ventilation
Measure: Count of Participants; unit: Participants
Arm/Group | MTPI Group | Classic Induction Group
Number analyzed (Participants) | 64 | 68
Participants | 62 | 66

3. Secondary Outcome: Number of Times Tracheal Intubations Are Attempted
Time Frame: after 5 minutes of successful ventilation
Measure: Count of Participants; unit: Participants
Arm/Group | MTPI Group | Classic Induction Group
Number analyzed (Participants) | 64 | 68
Participants
  1 time | 62 | 66
  2 times | 1 | 1
  3 times | 1 | 1

4. Secondary Outcome: Number of Participants for Whom Tracheal Intubations Failed
Time Frame: after 3 failed intubation attempts (less than 7 minutes from start of intubation)
Measure: Count of Participants; unit: Participants
Arm/Group | MTPI Group | Classic Induction Group
Number analyzed (Participants) | 64 | 68
Participants | 0 | 0

5. Secondary Outcome: Airway Cord View at the Time of Laryngoscopy as Categorized by the Modified Cormack-Lehane Classification (Before External Manipulation)
Description: The Cormack-Lehane classification system is a method used to categorize the airway view at the time of laryngoscopy. Data is reported categorically as follows 1(Full view of glottis),2(Partial view of glottis), 3(Only epiglottis seen, none of glottis seen) and 4(Neither glottis nor epiglottis seen)
Time Frame: from start of induction to 5 minutes of successful ventilation
Measure: Count of Participants; unit: Participants
Arm/Group | MTPI Group | Classic Induction Group
Number analyzed (Participants) | 64 | 68
Participants
  1 | 32 | 30
  2 | 32 | 34
  3 | 0 | 4
  4 | 0 | 0

6. Secondary Outcome: Minimum Systolic Blood Pressure
Time Frame: from the start of induction drug administration to about 5 minutes after successful ventilation
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | MTPI Group | Classic Induction Group
Number analyzed (Participants) | 64 | 68
mmHg | 130.6 (26.0) | 117.4 (24.5)

7. Secondary Outcome: Maximum Systolic Blood Pressure
Time Frame: from the start of induction drug administration to about 5 minutes after successful ventilation
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | MTPI Group | Classic Induction Group
Number analyzed (Participants) | 64 | 68
mmHg | 150.7 (21.6) | 145.3 (24.9)

8. Secondary Outcome: Minimum Diastolic Blood Pressure
Time Frame: from the start of induction drug administration to about 5 minutes after successful ventilation
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | MTPI Group | Classic Induction Group
Number analyzed (Participants) | 64 | 68
mmHg | 77.2 (17.1) | 69.4 (16.2)

9. Secondary Outcome: Maximum Diastolic Blood Pressure
Time Frame: from the start of induction drug administration to about 5 minutes after successful ventilation
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | MTPI Group | Classic Induction Group
Number analyzed (Participants) | 64 | 68
mmHg | 94.5 (18.1) | 92.0 (17.5)

10. Secondary Outcome: Minimum Heart Rate
Time Frame: from the start of induction drug administration to about 5 minutes after successful ventilation
Measure: Mean (Standard Deviation); unit: beats per minute (BPM)
Arm/Group | MTPI Group | Classic Induction Group
Number analyzed (Participants) | 64 | 68
beats per minute (BPM) | 77.3 (13.6) | 69.0 (13.5)

11. Secondary Outcome: Maximum Heart Rate
Time Frame: from the start of induction drug administration to about 5 minutes after successful ventilation
Measure: Mean (Standard Deviation); unit: beats per minute (BPM)
Arm/Group | MTPI Group | Classic Induction Group
Number analyzed (Participants) | 64 | 68
beats per minute (BPM) | 103.6 (17.7) | 103.0 (19.1)

12. Secondary Outcome: Minimum Oxygen Saturation (SpO2)
Time Frame: from the start of induction drug administration to about 5 minutes after successful ventilation
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | MTPI Group | Classic Induction Group
Number analyzed (Participants) | 64 | 68
Percentage | 95.3 (6.0) | 96.5 (4.4)

13. Secondary Outcome: Maximum Oxygen Saturation (SpO2)
Time Frame: from the start of induction drug administration to about 5 minutes after successful ventilation
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | MTPI Group | Classic Induction Group
Number analyzed (Participants) | 64 | 68
Percentage | 99.7 (0.6) | 99.8 (0.6)

14. Secondary Outcome: Expired Tidal Volume
Time Frame: from the start of induction drug administration to about 5 minutes after successful ventilation
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | MTPI Group | Classic Induction Group
Number analyzed (Participants) | 64 | 68
mL | 503.8 (84.0) | 507.3 (86.8)

15. Secondary Outcome: End-tidal Carbon Dioxide (CO2) Level
Time Frame: from the start of induction drug administration to about 5 minutes after successful ventilation
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | MTPI Group | Classic Induction Group
Number analyzed (Participants) | 64 | 68
mmHg | 32.2 (5.7) | 32.9 (6.4)

16. Secondary Outcome: Number of Participants That Had Injury Associated With Intubation
Description: Injury is defined as injury of teeth, lips, tongue, and pharyngeal bleed
Time Frame: within 24 hours after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | MTPI Group | Classic Induction Group
Number analyzed (Participants) | 64 | 68
Participants | 0 | 0

17. Secondary Outcome: Physical Response During Intubation, as Assessed by the Number of Participants Who Moved
Time Frame: during surgery
Measure: Count of Participants; unit: Participants
Arm/Group | MTPI Group | Classic Induction Group
Number analyzed (Participants) | 64 | 68
Participants | 0 | 2

18. Secondary Outcome: Physical Response During Intubation, as Assessed by the Number of Participants Who Coughed
Time Frame: during surgery
Measure: Count of Participants; unit: Participants
Arm/Group | MTPI Group | Classic Induction Group
Number analyzed (Participants) | 64 | 68
Participants | 0 | 0

19. Secondary Outcome: Number of Participants Who Had Awareness of Muscle Paralysis Before Loss of Consciousness as Assessed by the Post Anesthesia Care Unit Survey of Modified Time Principle Induction
Description: Awareness of Muscle Paralysis or Weakness before loss of consciousness was assessed by the Post Anesthesia Care Unit Survey of Modified Time Principle Induction through in person interviews to evaluate explicit and implicit recall. Number of Participants with Positive Explicit recall and Positive Implicit recall are reported.
  Explicit recall: Participants were asked, "Describe the last thing you remember before falling asleep." If the participant describes memories of paralysis or awareness of the intubation event this is classified as positive explicit recall. If none of these memories are described it is considered negative explicit recall.
  Implicit recall: Participants with negative explicit recall, were asked "Did you ever feel weakness or paralysis as you fell asleep?" If they answered yes, this is classified as positive implicit recall.
Time Frame: within one hour after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | MTPI Group | Classic Induction Group
Number analyzed (Participants) | 64 | 68
Participants
  Positive Explicit recall | 0 | 0
  Positive Implicit Recall | 2 | 3

20. Secondary Outcome: Level of Throat Soreness as Assessed by a Question on the Post Anesthesia Care Unit Survey of Modified Time Principle Induction
Description: Level of throats soreness is scored from 0(no pain) to 10(worst pain), a higher number indicating worse throat soreness.
Time Frame: within one hour after surgery
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MTPI Group | Classic Induction Group
Number analyzed (Participants) | 64 | 68
score on a scale | 3.3 (3.2) | 3.1 (2.8)

21. Secondary Outcome: Number of Participants Who Had Nausea as Assessed by the Post Anesthesia Care Unit Survey of Modified Time Principle Induction
Time Frame: within one hour after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | MTPI Group | Classic Induction Group
Number analyzed (Participants) | 64 | 68
Participants | 11 | 9

22. Secondary Outcome: Overall Patient Satisfaction as Assessed by a Question on the Post Anesthesia Care Unit Survey of Modified Time Principle Induction
Description: Patient satisfaction is scored from 0(not satisfied) to 10(extremely satisfied), a higher number indicating greater satisfaction.
Time Frame: within one hour after surgery
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MTPI Group | Classic Induction Group
Number analyzed (Participants) | 64 | 68
score on a scale | 9.3 (1.7) | 9.4 (0.9)

23. Secondary Outcome: Number of Participants Who Had Recollection of Pain on Induction
Time Frame: within one hour after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | MTPI Group | Classic Induction Group
Number analyzed (Participants) | 64 | 68
Participants | 4 | 0

24. Secondary Outcome: Provider Determination of Intubating Conditions, Based on Whether Intubation Was Classified as "Not Difficult" or "Difficult"
Time Frame: at time of surgery
Measure: Count of Participants; unit: Participants
Arm/Group | MTPI Group | Classic Induction Group
Number analyzed (Participants) | 64 | 68
Participants
  Difficult | 1 | 3
  Not Difficult | 63 | 65

25. Secondary Outcome: Number of Participants Who Had Vomiting as Assessed by the Post Anesthesia Care Unit Survey of Modified Time Principle Induction
Time Frame: within one hour after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | MTPI Group | Classic Induction Group
Number analyzed (Participants) | 64 | 68
Participants | 0 | 1

ADVERSE EVENTS:
Time Frame: Up to 24 hours
Arm/Group | MTPI Group | Classic Induction Group
All-Cause Mortality (participants affected / at risk) | 0/77 | 0/77
Serious Adverse Events (participants affected / at risk) | 0/77 | 0/77
Other Adverse Events (participants affected / at risk) | 0/77 | 0/77

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-01-28): https://cdn.clinicaltrials.gov/large-docs/92/NCT05509192/Prot_SAP_000.pdf